CLINICAL TRIAL: NCT05268900
Title: Effect of Different Ventilation Modes on Intracranial Pressure During Laparoscopic Colectomy Guided by Optic Nerve Sheath Diameter Measurement.
Brief Title: Ventilation Modes Effect on Intracranial Pressure During Laparoscopic Colectomy by Optic Nerve Sheath Diameter
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MD/ 21.10.553
Record Dates: First submitted 2022-01-26; First posted 2022-03-07 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-02

CONDITIONS: Laparoscopic Colectomy
Keywords: ventilation; intracranial pressure; laparoscopy
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Volume control ventilation group (Placebo Comparator): Patients' lungs will be ventilated with volume control ventilation mode
  Interventions: Device: Volume control ventilation group
- Pressure control ventilation-volume guaranteed group (Active Comparator): patients' lungs will be ventilated with Pressure control ventilation-volume guaranteed mode
  Interventions: Device: Pressure control ventilation-volume guaranteed group

INTERVENTIONS:
Device: Volume control ventilation group — Volume control ventilation mode
  Arms: Volume control ventilation group
Device: Pressure control ventilation-volume guaranteed group — Pressure control ventilation-volume guaranteed mode
  Arms: Pressure control ventilation-volume guaranteed group

SUMMARY:
Patients who undergo laparoscopic surgery often experience increased intracranial pressure (ICP). In laparoscopic colectomy surgery, the duration always exceeds 2h with more liability to changes in arterial blood gases, hemodynamics, also the patient is in Trendelenburg position about 30° head down, Trendelenburg position is believed to create changes in hemodynamics, respiratory mechanics, metabolic response, and ICP as it affects vital organs especially if steep positioning. Various modes of mechanical ventilation have been experimented to achieve good intraoperative oxygenation which may cause changes in arterial blood gas values and hemodynamic parameters that might lead to changes in the ICP. In this study we will measure ONSD, basal, intraoperative, and in the PACU to evaluate the effect of different ventilation modes (both VCV mode and PCV-VG mode) on intracranial pressure.

DETAILED DESCRIPTION:
The aim of the current study is to compare the effect of volume control ventilation (VCV) versus pressure control ventilation-volume guaranteed (PCV-VG) as modes of mechanical ventilation on ICP by US guided ONSD measurement during laparoscopic colectomy,

ELIGIBILITY:
Inclusion Criteria:

* Body mass index less than 30
* American Society of Anesthesiologist physical class I -III.

Exclusion Criteria:

* Patient refusal
* operative time < 2 hour (h)
* Patients with preexisting eye disease.
* History of eye surgery
* Optic nerve disease.
* Causes of elevated ICP.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Changes in ONSD O(optic) N(nerve) S(sheath) D(diameter) | Changes from baseline, till 30 minutes after recovery from anaesthesia
  ONSD is the acronym of O(optic) N(nerve) S(sheath) D(diameter), that ONSD is a non invasive method for measurement of intracranial pressure The optimal cutoff value has not been established, they vary between 4.85 and 5.9 mm and >5.9 mm is a sure sign of increased intracranial tension

SECONDARY OUTCOMES:
Heart rate | Changes from baseline, till 30 minutes after recovery from anaesthesia
  is allowed to swing within 20% of the basal value
Mean arterial blood pressure | Changes from baseline, till 30 minutes after recovery from anaesthesia
  is allowed to swing within 20% of the basal value
Peak airway pressure | intra-operative changes from time of induction of anesthesia and intubation (post induction), till the end of surgery (before extubation).
  Peak airway pressure values should not exceed 30 cm H2O. Values greater than 40 cm H2O may be harmful to the normal lung. Peak pressure applies when there is airflow in the circuit, i.e.the maximum pressure during inspiration . What determines the peak pressure is the airway resistance in the lungs. So if there is a problem with the airways the peak pressure will rise.
Plateau airway pressure | intra-operative changes from time of induction of anesthesia and intubation (post induction), till the end of surgery (before extubation).
  Plateau pressure is the pressure applied to small airways and alveoli during positive-pressure mechanical ventilation.when there is no air flow in the circuit. That is when inspiration is complete. This pressure is determined by the lung compliance. So it follows that if there is a problem with the compliance the plateau pressure will rise.
  Plateau pressure is measured during an inspiratory pause on the mechanical ventilator.
  Pplat is never bigger than PIP and is typically <10 cm H2O lower than PIP when airway resistance is not elevated.
mean airway pressure | intra-operative changes from time of induction of anesthesia and intubation (post induction), till the end of surgery (before extubation).
  mean airway pressure typically refers to the mean pressure applied during positive-pressure mechanical ventilation. Mean airway pressure correlates with alveolar ventilation, arterial oxygenation, hemodynamic performance, and barotrauma
Dynamic Lung compliance | intra-operative changes from time of induction of anesthesia and intubation (post induction), till the end of surgery (before extubation).
  dynamic lung compliance Cdyn = VT / (PIP - PEEP)…..change in volume/change in pressure, where airflow resistance becomes a factor. which ranges physiologically in adults between 50 - 80 ml/cm H2O while for intubated, mechanically ventilated adults is about 30 to 40 ml/cm H2O
Static Lung compliance | intra-operative changes from (post induction) just after induction of anesthesia and intubation, till the end of surgery (before extubation).
  static compliance and dynamic compliance static lung compliance....Cstat = VT/ ( Pplat - PEEP) ….change in volume/change in pressure when there is no air flow..... The physiological Cstat for adult is 70 - 100 while for intubated, mechanically ventilated adults is about 50 to 60 ml/cm H2O
pH | Changes from baseline, till 30 min after recovery from anesthesia.
  PH ranges normally between 7.35 - 7.45 when >7.45 it is alkalosis when <7.35 it is acidosis
PaCO2 (carbon dioxide tension) | Changes from baseline, till 30 min after recovery from anesthesia.
  PaCo2 which ranges normally between 35 -45 mmHg it increase above 45 with causes of hypercapnia as hypoventilation and insufflation with Co2 and decrease below 35 with hypotension, hypo-perfusion and excessive hyperventilation Normal PaCO2-EtCO2 difference is 2-5 mmHg
Headache | for 24 hour after surgery
  the severity of headache will be recorded using visual analogue score (where 0 = no pain and 10 = worst pain imaginable), mild headache pain will be defined by scores 1-4, moderate; by scores 5-7, and severe; by scores 8-10.
Postoperative nausea and vomiting | for 24 hour after surgery
  Nausea will be explained to all patients, where ( 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms, 3 = severe symptoms ) and also the incidence of vomiting will be recorded by asking a questionnaire to all patients; is vomiting present or absent.
PaO2 (partial pressure of arterial oxygen) | Changes from baseline, till 30 min after recovery from anesthesia
  PaO2 should= FiO2 x 500 (e.g. 0.21 x 500 = 105 mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Hanaa M El Bendary, Study Director — Assistant professor, MD anesthesia Department, Faculty of Medicine,; Doaa G Diab, Study Chair — professor, MD anesthesia Department, Faculty of Medicine, Mansoura University, Egypt
Locations (1):
- Mansoura University, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Deidentiﬁed individual participant data for all primary and secondary outcome measures will be made available
Supporting Information: SAP, ICF, CSR, Analytic Code
Time Frame: will be available within 6 months of study completion
Access Criteria: data access requests will be reviewed by an external independent review panel. requestors will be required to sign a data access agreement